CLINICAL TRIAL: NCT04215861
Title: Clinical Study on Raman Spectra of Blood, Saliva and Urine in Patients With Cancer Treated by Modern Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PJ-KS-KY-2019-135
Record Dates: First submitted 2019-12-11; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer; Liver Cancer; Stomach Cancer; Breast Cancer
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms; Stomach Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood, saliva and urine samples of tumor patients on the day of admission and discharge were collected for Raman spectral analysis, which provided exploration for the prediction of efficacy, follow-up and prognosis according to the variation characteristics of Raman spectral.

DETAILED DESCRIPTION:
Blood, saliva and urine samples of tumor patients on the day of admission and discharge were collected for Raman spectral analysis, which provided exploration for the prediction of efficacy, follow-up and prognosis according to the variation characteristics of Raman spectral

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* The patient whose tumor (tissue or cell) was first diagnosed by pathology;
* Plan to receive routine clinical treatment: chemotherapy, radiotherapy, surgery, intervention, targeted therapy, traditional Chinese medicine treatment and biological immunotherapy;
* Have relevant indications for treatment and have no contraindications;

Exclusion Criteria:

* Severe or uncontrollable systemic diseases (such as unstable or uncompensated respiratory, heart, liver or kidney diseases, etc.);
* Other circumstances considered inappropriate by the researcher to participate in the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 18-80 years old;
  * The patient whose tumor (tissue or cell) was first diagnosed by pathology;
  * Plan to receive routine clinical treatment: chemotherapy, radiotherapy, surgery, intervention, targeted therapy, traditional Chinese medicine treatment and biological immunotherapy;
  * Have relevant indications for treatment and have no contraindications;
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Raman spectra | the 1st day before operation
  Blood, saliva and urine samples of tumor patients on the day of admission and discharge were collected to analyze the signal changes of Raman spectrum
Raman spectra | the 1st day after operation
  Blood, saliva and urine samples of tumor patients on the day of admission and discharge were collected to analyze the signal changes of Raman spectrum

SECONDARY OUTCOMES:
progression-free survival | through study completion, an average of 1 year
overall survival | through study completion, an average of 1 year
objective response rate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD,PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided